CLINICAL TRIAL: NCT04010266
Title: Safety and Effectiveness of Virtual Reality Utilizing RelieVRx for Total Knee Arthroplasty (TKA) for the Reduction of Acute Postoperative Pain and Opioid Use
Brief Title: RelieVRx for Total Knee Arthroplasty (TKA) for the Reduction of Acute Postoperative Pain and Opioid Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AppliedVR Inc. (Industry)
Collaborators: Geisinger Clinic (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-0388; 2R44DA049640 (NIH)
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Opioid Use; Arthropathy of Knee; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care group (Active Comparator): Receive standard of care for pain management, do not receive RelieVRx headset
  Interventions: Drug: multi-modality pain management
- Standard of care + RelieVRx group (Experimental): Receive standard of care for pain management, plus RelieVRx headset
  Interventions: Device: RelieVRx headset; Drug: multi-modality pain management

INTERVENTIONS:
Device: RelieVRx headset — RelieVRx is a virtual reality therapy intended as adjunctive treatment for acute surgical pain
  Arms: Standard of care + RelieVRx group
Drug: multi-modality pain management — combination of medications may be used such as a local anesthesia, ibuprofen, acetaminophen, gabapentin, ketamine, lidocaine, and opioids

SUMMARY:
This is a single-center, prospective, randomized, controlled study of the appliedVR RelieVRx headset in subjects undergoing Total Knee Arthroplasty (TKA). This study will evaluate two primary endpoints - effectiveness of a single use of RelieVRx in the reduction of acute postoperative pain by 20%; and overall effectiveness of RelieVRx as an opioid-sparing intervention, where opioid consumption is reduced by at least 20% over a 90-day postoperative period in the interventional, standard of care (SOC) plus RelieVRx group compared to the control, SOC group.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, controlled study of the appliedVR RelieVRx headset in subjects undergoing Total Knee Arthroplasty (TKA). Patients will be randomized to one of the two groups after study enrollment, and patients in the test arm will be educated about the device preoperatively to facilitate its use in the acute post-operative period. The goals of VR will be presented in the context of an alternate method of pain control to opioids. This study will evaluate two primary endpoints - effectiveness of a single use of RelieVRx in the reduction of acute postoperative pain by 20%; and overall effectiveness of RelieVRx as an opioid-sparing intervention, where opioid consumption is reduced by at least 20% over a 90-day postoperative period in the interventional, standard of care (SOC) plus RelieVRx group compared to the control, SOC group.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old
2. Subject is willing and able to read, comprehend, and sign the study informed consent form in English prior to study specific procedure
3. Subject is scheduled for Total Knee Arthroplasty (TKA) surgery
4. Subject has a score of 1-3 based on the American Society of Anesthesiologists Physical Status Classification System
5. Subject attended the pre-op Total Joint Arthroplasty Patient Education class (Proven Recovery Program©)
6. Subject agrees to be enrolled in Force Therapeutics, a web-based, digital rehabilitation and education program
7. Subject has family member or community support during post-surgical recovery period

Exclusion Criteria:

1. Diagnosed with chronic pain syndrome
2. Body Mass Index (BMI) ≥ 40
3. Current tobacco user at time of surgery
4. Uncontrolled sleep apnea
5. Bilateral TKA
6. Current or recent history (in past year) of substance abuse disorder
7. Uncontrolled diabetes (HbA1c ≥ 7.0) 7.8 at time of surgery
8. History of Pulmonary Embolism (PE) or Deep Vein Thrombosis (DVT)
9. Currently being treated with blood thinners at time of surgery
10. Diagnosis of Rheumatoid Arthritis (RA)
11. Has Methicillin-resistant Staphylococcus aureus (MRSA)
12. Currently pregnant/breastfeeding or planning to in the next 3 months
13. Comorbidities including neurological, psychosocial, sensory, or other disorders that may impact pain perception
14. Diagnosis of epilepsy, dementia, migraines, or other neurological disorders that may prevent VR usage, and/or other medical conditions predisposed to nausea and dizziness
15. Hypersensitivity to flashing lights or motion
16. Claustrophobia
17. Lack of stereoscopic vision
18. Severe hearing impairment
19. Injury to eyes, face, or neck that prevents comfortable VR usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Suk, Principal Investigator — Geisinger Clinic
Locations (3):
- United States (3):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Geisinger South Wilkes Barre, Wilkes-Barre, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Group | Standard of Care + RelieVRx Group
Started | 32 | 31
Completed | 24 | 18
Not Completed | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Group | Standard of Care + RelieVRx Group | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (12.5) | 51.4 (13.8) | 50.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 17 | 17 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 30 | 29 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Numerical Pain Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Rating make on a scale from 0 to 10 where 0 implies no pain and 10 implies pain that is unbearable. Thus, increasing values of the Numerical Pain Rating Scale imply greater amounts of pain
  units on a scale | 5.78 (1.54) | 5.76 (1.34) | 5.77 (1.44)

OUTCOME MEASURES:

1. Primary Outcome: Acute Postoperative Pain
Description: Visual Analog Pain scale; worst 0-10 best
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care Group | Standard of Care + RelieVRx Group
Number analyzed (Participants) | 32 | 31
units on a scale | 5.13 (1.79) | 4.42 (1.17)

2. Primary Outcome: Opioid Consumption
Description: Morphine Milligram Equivalents (MME)
Time Frame: 90 days
Population: Morphine milligram equivalents were measured preoperatively and postoperatively for each patient. The outcome measure reported is the median change in total MME from pre-op to Post-op
Measure: Median (Inter-Quartile Range); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Standard of Care Group | Standard of Care + RelieVRx Group
Number analyzed (Participants) | 24 | 18
Morphine Milligram Equivalents (MME) | -28.0 [-35.0 to -23.5] | -34.8 [-37.0 to -23.5]

3. Secondary Outcome: KOOS Jr. Score
Description: short form of knee injury and osteoarthritis outcome score; worst 0 - 100 best
Time Frame: 90 days
Population: Change in KOOS Jr from Pre-surgery to post-surgery, median (IQR)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care Group | Standard of Care + RelieVRx Group
Number analyzed (Participants) | 24 | 18
score on a scale | 27.6 [17.5 to 38.0] | 32.2 [21.2 to 42.0]

4. Secondary Outcome: Veterans RAND 12 Health Survey (VR-12) - Physical Component Score
Description: This is a measure of quality of life. The VR-12 provides a physical component score (i.e., physical health domain) that provides larger weights for four of the domains (physical function, role-physical, bodily pain, and general health). This is a 12 items survey. VR-12 scores are standardized using a T-score metric with a mean of 50 and a standard deviation of 10. Larger values imply greater physical function and quality of life.
Time Frame: 90 days
Population: Change in VR-12 from Pre-surgery to post-surgery, median (IQR)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care Group | Standard of Care + RelieVRx Group
Number analyzed (Participants) | 24 | 18
score on a scale | 7.2 [2.0 to 11.4] | 9.5 [4.0 to 12.8]

ADVERSE EVENTS:
Time Frame: 4 months for each patient
Arm/Group | Standard of Care Group | Standard of Care + RelieVRx Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT04010266/Prot_SAP_000.pdf